CLINICAL TRIAL: NCT06732024
Title: Using Vaccum Assisted Closure of Wound Instead of Primary Closure As Prophylactic Way Against Burst Abdomen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Hassan Anwar Ali, resident doctor at general surgery department Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Vaccum/primary closure burst
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Burst Abdomen
Keywords: Vaccum Assisted Closure; primary closure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): Vaccum Assisted Closure of Wound
  Interventions: Procedure: Vaccum assisted closure
- group B (Experimental): primary closure Closure of Wound
  Interventions: Procedure: primary wound closure

INTERVENTIONS:
Procedure: Vaccum assisted closure — close skin and SC tissue by vaccum device
  Arms: group A
Procedure: primary wound closure — close skin and SC tissue by primary closure
  Arms: group B

SUMMARY:
A vacuum-assisted closure (VAC) device also known as negative pressure wound therapy (NPWT), is a medical treatment used to promote wound healing, it involves using a specialized device to apply negative pressure (suction) to a wound, which helps to accelerate the healing process.

Benefits :

Improved Healing: By removing excess fluid and reducing edema, the VAC device promotes faster wound healing and tissue repair.

Reduced Risk of Infection: The negative pressure helps to reduce bacterial load and create a more favorable environment for healing.

Enhanced Perfusion: The suction can improve blood flow to the wound area, aiding in the delivery of nutrients and oxygen essential for healing.

Granulation Tissue Formation: The therapy encourages the growth of new tissue (granulation tissue) which fills the wound and supports closure.

Overall, VAC therapy is a valuable tool in modern wound care, particularly for complex or difficult-to-heal wounds. If you or someone you know is considering or using this therapy, it's important to follow the guidance of healthcare professionals to maximize its effectiveness and manage any potential risks.

the study aim to evaluate patients , identify high risk ones , preparing to close wound of laparotomy with vaccum assisted device instead of primary closure with suturing till patient's general condition improve then delayed primary closure and comparing that to high risk patients who close wound primarily with suturing in terms of rate of burst abdomen …this is a randomized controlled trial

DETAILED DESCRIPTION:
Burst abdomen (abdominal wound dehiscence) is a severe post-operative complication. Incidence as described in literature ranges from 0.4% to 3.5% … Burst abdomen is defined as post-operative separation of abdominal Musculo-aponeurotic layers, which is recognized within days after surgery and requires some form of intervention. Various risk factors are responsible for wound dehiscence such as emergency surgery, intra-abdominal infection, malnutrition (hypoalbuminemia, anemia), advanced age, systemic diseases (uremia, diabetes mellitus) etc…. Good knowledge of these risk factors is mandatory for prophylaxis… Patient identified as being high risk may benefit from close observation and early intervention

ELIGIBILITY:
Inclusion Criteria:

* intraabdominal sepsis (wbc:>12000,HR>90,T>38,tachypnea and proven infection) Malnutrition including anaemia and hypoproteinemia Chronic diseases including diabetes and uremia Increased intra abdominal pressure including persistent coughing ,diffuse gaseous distention Smoking Previous abdominal surgery Old age Steroid use

operation : Emergency not elective ones Dirty or contaminated Those involving colostomy and ileostomy that is close to wound

Exclusion Criteria:

* Patients having elective surgery Absence of intra abdominal sepsis Negative exploration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative burst abdomen in both group | 1 month
  number of patients who will have burst abdomen after surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Waqar SH, Malik ZI, Razzaq A, Abdullah MT, Shaima A, Zahid MA. Frequency and risk factors for wound dehiscence/burst abdomen in midline laparotomies. J Ayub Med Coll Abbottabad. 2005 Oct-Dec;17(4):70-3. PMID 16599042